CLINICAL TRIAL: NCT00241787
Title: Progression of Sub-Clinical Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1314; R01HL081352 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Carotid Artery Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To determine the rate of progression of sub-clinical cardiovascular disease as measured in carotid intimal medial thickness over a period of 8 to 10 years.

DETAILED DESCRIPTION:
BACKGROUND:

Strong associations exist between cardiovascular events and increased carotid artery wall intima-media thickness (IMT) as measured non-invasively by carotid ultrasound. Carotid IMT is accepted as a surrogate marker of sub-clinical cardiovascular disease.The study will determine the rate of progression of sub-clinical cardiovascular disease (change in IMT) over a period of 8 to 10 years.

DESIGN NARRATIVE:

The study will determine the rate of progression of sub-clinical cardiovascular disease (change in intimal medial thickness {IMT}) over a period of 8 to 10 years. Imaging and IMT measurements of approximately 2800 to 3000 members of the Framingham Offspring cohort having had baseline IMT measurements at their 1995-98 clinic visit will be repeated in 2005-2007. The principal aims of the project are to study the primary hypotheses that: 1. Interim exposure to traditional cardiovascular risk factors measured over 50 years is positively associated with the progression rate of carotid IMT. 2. Baseline carotid IMT and cumulative exposure to cardiovascular risk factors 20 years before the baseline visit are a better predictor of progression of sub-clinical disease after 8 to 10 years than the interim exposure to risk factors. 3. Novel risk factors such as C-reactive protein and homocysteine affect progression of carotid atherosclerosis more than traditional risk factors. This study will add a phenotypic marker of site-specific change in sub-clinical cardiovascular disease to the Framingham Study database. This complements ongoing research on the progression of sub-clinical cardiovascular disease and its associations with family history of premature cardiovascular events and genomic markers

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community based in Framingham MA
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Actual)
Dates: Start 2005-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Morbidity | Longitudinal follow-up
  Longitudinal follow-up of community based cohort

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Polak, MD, MPH, Principal Investigator — Tufts Medical Center